CLINICAL TRIAL: NCT05061407
Title: An African, International Multi-centre Fourteen-day Evaluation of Patient Care and Clinical Outcomes for Paediatric Patients Undergoing Surgery (ASOS-Paeds)
Brief Title: An African, Multi-centre Evaluation of Patient Care and Clinical Outcomes for Paediatric Patients Undergoing Surgery
Acronym: ASOS-Paeds
Status: Completed | Type: Observational
Sponsor: University of KwaZulu (Other)
Collaborators: University of Cape Town (Other); African Perioperative Research Group (APORG) (Unknown); Safe Surgery South Africa (SSSA) (Unknown)
Responsible Party: Principal Investigator, Alexandra Torborg, Principal Investigator, University of KwaZulu
Other Study IDs: ASOS-Paeds
Record Dates: First submitted 2021-09-04; First posted 2021-09-29 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Paediatric Surgery; Perioperative/Postoperative Complications; Perioperative Outcomes; Hospital Mortality; Developing Countries; Outcome Assessment; Paediatrics; Prospective Studies; Surgery
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paediatric surgical patients: All patients < 18 years old, admitted to participating hospitals during the study period who undergo elective and non-elective surgery

SUMMARY:
Access to safe surgery is a basic human right. This is highlighted by the work of the Lancet Commission on Global Surgery. There is a large burden of surgical disease in the paediatric surgical population with a large unmet need. In Africa, children comprise a significant proportion of the population with approximately 50% of the population being ≤19 years old. Limited data from Africa suggests the risk factors for, incidence and outcomes associated with paediatric surgical complications differ from HICs.

The African Surgical Outcomes Study (ASOS) has described surgical outcomes in adult patients in Africa.

There is a need to determine the burden of the complications in paediatric surgical patients in Africa, and the risk factors for and the type of complications experienced. Once this study is completed, the investigators will be able to target appropriate interventions to improve surgical outcomes for children in Africa. The investigators have the capacity to do this important work, through the African Perioperative Research Group (APORG) group.

DETAILED DESCRIPTION:
Surgery is a cost-effective public health intervention. There are significant disparities in access to and the safety of surgical and anaesthesia services in low and middle-income countries (LMICs) compared to high-income countries (HICs). There is a large burden of surgical disease in the paediatric surgical population with a large unmet need. In Africa, children comprise a significant proportion of the population with approximately 50% of the population being ≤19 years old.

Postoperative complications are an important determinant of surgical morbidity and mortality. Limited data from Africa suggests the risk factors for, incidence and outcomes associated with paediatric surgical complications differ from HICs. In the prospective, observational South African Paediatric Surgical Outcomes Study (SAPSOS), the patients in this middle-income country (MIC), had double the incidence of complications, and the types of complications differed from HICs, with a predominance of infective complications. Furthermore, the risk factors for complications (ASA physical status, urgency of surgery, severity of surgery and infective indication for surgery) were different from HICs, where risk factors include gestational age, ASA physical status >3, a history of cardiovascular disease, and cardiovascular, neurological, or orthopaedic surgical procedures. Postoperative mortality was ten times higher in South Africa than in a prospective study in HICs. A prospective study of paediatric perioperative mortality in 24 Kenyan hospitals showed a 7 day postoperative mortality of 1.7%, which is 17 times higher than that reported in HICs.

The African Surgical Outcomes Study (ASOS) has described surgical outcomes in adult patients in Africa. Patients had a lower risk profile and fewer complications compared to those in HICs. However, the postoperative mortality was twice that of the global average.

There is a need to determine the burden of the complications in paediatric surgical patients in Africa, and the risk factors for and the type of complications experienced. Once this study is completed, the investigators will be able to target appropriate interventions to improve surgical outcomes for children in Africa. The investigators have the capacity to do this important work, through the African Perioperative Research Group (APORG) group.

STUDY OBJECTIVE To determine the incidence of in-hospital postoperative complications up to 30 days post-surgery in paediatric surgical patients <18 years in Africa

STUDY DESIGN Fourteen-day, international African multi-centre prospective cohort study of paediatric patients (<18 years) undergoing surgery. This study will be registered on ClinicalTrials.gov. Patients will be followed up for a maximum of 30 days.

The primary outcome is the incidence of in-hospital postoperative complications in paediatric surgical patients in Africa. Secondary outcome measures include mortality rate for patients < 18 years undergoing surgery in Africa, risk factors associated with in-hospital complications, time from first presentation to operation, incidence of severe intraoperative critical incidents, level of qualification of anesthesia and surgery providers and number of specialists per paediatric population, and rate of admission to critical care.

The intention is to present a representative sample of paediatric surgical outcomes across all African countries. This study will run from October 2021 until December 2022.

ETHICS APPROVAL A waiver of consent has been approved by the IRB with the proviso that an approved broadcasting document and pictorial description are both placed for patients to see around the hospital and in the relevant wards. The requirement for patient consent is expected to vary according to regulations of the participating nations. the national leaders will ensure ethics approval is obtained form their respective countries and centres. Centres will not be permitted to record data unless ethics approval and an equivalent waiver is in place.

PREPARATORY WORK Prior leadership in the South African Paediatric Surgical Outcomes Study (SAPSOS) and the African Surgical Outcomes Study (ASOS) have ensured tested resource resources necessary to run this study. This will be the first continental collaborative study of paediatric surgical outcomes in Africa.

IMPORTANCE OF THIS STUDY Surgery is associated with significant morbidity. Accurate information regarding the burden of morbidity and mortality associated with paediatric surgery in Africa would allow for appropriate allocation of resources in the future, and the implementation of interventions to improve paediatric patient outcomes. This study therefore has important public health implications for Africa. This study will also provide the necessary data to develop future collaborative work to improve African surgical paediatric patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients < 18 years, admitted to participating hospitals during the study period
* elective and non-elective surgery (including day case surgery)
* operative procedures outside operating theatres where a general anaesthetic (GA) is performed.

Exclusion Criteria:

1. radiological or other procedures not requiring general anaesthesia, or where general anaesthesia is performed but no procedure is performed e.g. general anaesthesia during magnetic resonance imaging (MRI).
2. Obstetric surgery.
3. Prior participation in ASOS-Paeds.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients less than 18 years old, admitted to participating hospitals during the study period who undergo elective and non-elective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 8625 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | Until hospital discharge censored at 30 days postoperative
  Incidence of in-hospital postoperative complications in paediatric surgical patients in Africa.

SECONDARY OUTCOMES:
Postoperative mortality | Until hospital discharge censored at 30 days postoperative
  1 a. The day of surgery mortality rate for patients < 18 years undergoing surgery in Africa.
  b. The in-hospital mortality rate for patients < 18 years undergoing surgery in Africa censored at 30 days.
Access to surgery | Until hospital discharge censored at 30 days postoperative
  Time from first presentation to operation
Intraoperative critical incidents | Until hospital discharge censored at 30 days postoperative
  Incidence of severe intraoperative critical incidents
Anesthesia and surgery providers | Until hospital discharge censored at 30 days postoperative
  Number of non-physician, nurse, physician (non-specialist), physician (specialist) anaesthesia and surgery providers
Rate of admission to critical care | Until hospital discharge censored at 30 days postoperative
  Percentage of patients requiring admission to critical care immediately postoperatively
Number of specialists per paediatric population | Within 6 months of the start of recruitment
  Number of specialists per paediatric population

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Torborg, Principal Investigator — University of KwaZulu
Locations (2):
- Inkosi Albert Luthuli Central Hospital, Durban, KwaZuluNatal, South Africa
- Ribat Teaching Hospital, Khartoum, Sudan

REFERENCES:
- [Derived] ASOS-Paeds Investigators. Outcomes after surgery for children in Africa (ASOS-Paeds): a 14-day prospective observational cohort study. Lancet. 2024 Apr 13;403(10435):1482-1492. doi: 10.1016/S0140-6736(24)00103-X. Epub 2024 Mar 22. PMID 38527482

DOCUMENTS (4):
  • Study Protocol (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/07/NCT05061407/Prot_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan ASOS-Paeds (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT05061407/SAP_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan Substudy Facilities (2024-09-03): https://cdn.clinicaltrials.gov/large-docs/07/NCT05061407/SAP_002.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan Severe Critical Events (2025-03-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT05061407/SAP_003.pdf